CLINICAL TRIAL: NCT03718923
Title: The Seaver Autism Center for Research and Treatment - Assessment Core
Brief Title: FOXP1 Syndrome: The Seaver Autism Center for Research and Treatment is Characterizing FOXP1-related Neurodevelopmental Disorders Using Genetic, Medical, and Neuropsychological Measures.
Status: Recruiting | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: The Seaver Foundation (Unknown); Autism Science Foundation (Other); Research Foundation for Mental Hygiene, Inc. (Other)
Responsible Party: Principal Investigator, Alexander Kolevzon, Clinical Director of the Seaver Autism Center for Research and Treatment, Professor of Psychiatry and Pediatrics and Director of Child and Adolescent Psychiatry, Icahn School of Medicine at Mount Sinai
Other Study IDs: GCO 98-436 - A
Record Dates: First submitted 2018-10-23; First posted 2018-10-25 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: FOXP1; Mental Retardation With Language Impairment and With or Without Autistic Features; Autism Spectrum Disorder
Keywords: FOXP1; Intellectual Disability; Autism Spectrum Disorder; Global Developmental Delay; Neurodevelopmental Deficits; Developmental Disability
MeSH Terms: conditions — Autism Spectrum Disorder; Intellectual Disability; Learning Disabilities; Developmental Disabilities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood and/or saliva samples from research participants who consent to giving biological specimens for research genetics may be retained with potential for extraction of DNA. Blood samples may be used to create Induced Pluripotent Stem Cells (iPSCs).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
FOXP1, also known as Forkhead-box Protein P1, is a transcription factor protein belonging to the FOX gene family. Disruptions in the FOXP1 gene cause a phenotype characterized by global developmental delay, speech deficits, mild dysmorphic features, and traits of autism spectrum disorder. This study seeks to characterize FOXP1-related neurodevelopmental disorders using a number of genetic, medical and neuropsychological measures.

DETAILED DESCRIPTION:
Subjects with a variant in the FOXP1 gene will be asked to complete a battery of developmental, behavioral and medical assessments to better characterize gene-related neurodevelopmental deficits. This series of assessments takes place over the course of a three-day period. It includes the Autism Diagnostic Observation Schedule (ADOS), parent interviews regarding developmental history and behavior, a psychiatric evaluation, a neurology assessment, as well as a clinical genetic evaluation that includes a physical and vitals exam. Affected individuals, as well as biologically related siblings, will also undergo a series of sensory assessments, including a research EEG, visual evoked potential, and an eyetracking assessment. Family members present for the visit will also be asked to provide a blood and/or saliva sample for research genetics.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants must have a documented variant affecting the FOXP1 gene that the research team determines to be likely or definitely pathogenic.
* Eligible participants must be at least 2 years of age.

Exclusion Criteria:

* none

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals for this cohort study will be selected from any population, provided that they have a variant in the FOXP1 gene and meet eligibility requirements.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2016-03-28 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Autism Diagnostic Observation Schedule (ADOS) | Day 1
  The ADOS is a structured, play-based assessment of communication, social interaction and behavior in individuals (children and adults) suspected of having a diagnosis of Autism Spectrum Disorder. The examiner will select 1 of 4 different ADOS modules, which differ based on chronological age and verbal fluency, to use for the individual being assessed. An Overall Total score >= 16, if the individual meets for the "few to no words" algorithm, or 12, if the individual meets for the "some words" algorithm, suggests autism in the individual. An Overall Total score of 11 to 15, if the individual meets for the "few to no words" algorithm, or 8 to 11, if the individual meets for the "some words" algorithm, suggests the individual is on the autism spectrum. An Overall Total score equal to or lower than 10, if the individual meets for "few to no words" algorithm, or 7, if the individual meets for the "some words" algorithm, classifies the individual as "non-spectrum" or not on the spectrum.

SECONDARY OUTCOMES:
Autism Diagnostic Interview - Revised (ADI-R) | Day 1
  The ADI-R is a standardized, semi-structured clinical assessment used to diagnose Autism Spectrum Disorder (ASD) in children and adults. The ADI-R is a structured interview administered by an examiner to the primary caregiver of children and adults suspected of having ASD. The assessment contains 93 items, scored from 0 (behavior not present) to 279 (severe or frequent behavior), A higher assessment score indicates poorer outcomes.
Stanford-Binet Intelligence Scales | Day 1
  The Stanford-Binet Intelligence Scales are a cognitive assessment measuring the five factors of fluid reasoning, knowledge, quantitative reasoning, visual-spatial processing and working memory. The number of correct responses for the subtests is converted to a Standard Age Score, based on the chronological age of the individual being assessed. The Area Scores and Test Composite on the Stanford-Binet test have an average score of 100 and a standard deviation of 16. The converted score of the individual being assessed indicates where he/she is relative to the norm. A score exceeding 145 is classified as "Genius or near genius," and scores below 70 are classified as "Borderline deficiency."
Differential Ability Scales (DAS) | Day 1
  The DAS is a battery of cognitive and achievement testing for children 2.5-18 years old that is divided into Early Years and School-Age versions. The 20 subtests of the DAS are broken up into 17 cognitive and 3 achievement subtests. The scores of the test are categorized into i) General Conceptual Ability (GCA) which is based on the ability of the individual being assessed to perform complex mental processing involving transformation of information ii) cluster scores that indicate verbal, spatial and nonverbal reasoning abilities and iii) subtest scores that represent specific abilities or processes. The tests yield t-scores and percentiles by age.
Mullen Scales of Early Learning | Day 1
  The Mullen Scales of Early Learning are a clinical assessment used to measure cognitive ability and motor development in children ages 0-68 months on the five scales of Gross Motor, Visual Reception, Fine Motor, Expressive Language, and Receptive Language. T-scores, percentile rankings, and age equivalents can be calculated for each of these five scales.

CONTACTS AND LOCATIONS:
Overall Officials: Elodie Drapeau, Ph.D., Principal Investigator — Icahn School of Medicine at Mount Sinai; Paige Siper, Ph.D., Principal Investigator — Icahn School of Medicine at Mount Sinai; Reymundo Lozano, M.D., Principal Investigator — Icahn School of Medicine at Mount Sinai; Alexander Kolevzon, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- The Seaver Autism Center for Research and Treatment, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No